CLINICAL TRIAL: NCT02943980
Title: Influenced the Type of Laryngoscopy the Intraoperative Nerve Monitoring During Thyroid Surgery; a Controlled, Randomized Study (LiON-Study)
Brief Title: Influenced the Type of Laryngoscopy the Intraoperative Nerve Monitoring During Thyroid Surgery
Acronym: LiON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Marc Kriege, MD, MD, Johannes Gutenberg University Mainz
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JGU
Record Dates: First submitted 2016-10-13; First posted 2016-10-25 (Estimated); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Thyroid; Airway Morbidity
Keywords: Intraoperative nerve monitoring, airway management
MeSH Terms: conditions — Thyroid Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CMAC Videolaryngoscope (Experimental): tracheal intubation using CMAC
  Interventions: Device: CMAC Videolaryngoscope
- Macintosh laryngoscope (Experimental): tracheal intubation using Macintosh laryngoscope
  Interventions: Device: Macintosh Laryngoscope

INTERVENTIONS:
Device: CMAC Videolaryngoscope — In a randomised order we evaluate the quality of the IONM after securing the airway with the CMAC
  Arms: CMAC Videolaryngoscope
Device: Macintosh Laryngoscope — In a randomised order we evaluate the quality of the IONM after securing the airway with the conventional Macintosh Laryngoscope
  Arms: Macintosh laryngoscope

SUMMARY:
A randomized controlled prospective study of laryngoscopy and evaluation of the Intraoperative nerve monitoring during thyroid surgery comparing direct laryngoscopy and the C-MAC videolaryngoscope.

DETAILED DESCRIPTION:
Intraoperative nerve monitoring (IONM) is used in addition to the visual the nerve in thyroid surgery. Here, the IONM can be done by placing electrodes on an endotracheal tube. In order to guarantee a sufficient signal quality of the IONM, the electrode must be adequately positioned on the glottis. The present study pursued the question of whether the conventional direct laryngoscopy compared with video laryngoscopy allows a visually adequate tube placement.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 Years No concurrent participation in another study
* capacity to consent
* Present written informed consent of the research participant
* Elective surgery under general anesthesia

Exclusion Criteria:

* Age <18 years
* Existing pregnancy
* Lack of consent
* inability to consent
* emergency patients
* Emergency situations in the context of a Difficult Airway Management
* ASA classification 4
* situations where the possibility of accumulated gastric contents
* Participation in another study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2017-01-03 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2019-02-15 (Actual)

PRIMARY OUTCOMES:
Evaluation of the quality of the IONM during thyroid surgery | Quality IONM; intraoperative 1-3 hours
  Evaluation of intraoperative loss of the EMG-Signal (Quality character of the IONM)

SECONDARY OUTCOMES:
intubation success | at intubation; < 120 Seconds
  successful tracheal intubation at the first attempt, compared to more than one attempt
Cormack and Lehane Classification | during the laryngoscopy; < 120 Seconds
  airway visualization during intubation process
Percentage of glottic opening | during the laryngoscopy; < 120 Seconds
  airway visualization during intubation process
IDS (intubation difficult score) | < 120 Seconds
  Summation of specific characters during the tracheal intubation

CONTACTS AND LOCATIONS:
Overall Officials: Marc Kriege, MD, Principal Investigator — University Medical Center
Locations (1):
- Department of Anesthesiology,Prof. C. Werner, Universitätsmedizin of the JG University, Mainz, Rhineland-Palatinate, Germany

IPD SHARING:
Plan to Share IPD: No